CLINICAL TRIAL: NCT03906955
Title: Testing a Brief, Theory-guided Video Chat Intervention for Enhancing Self-efficacy and Lifestyle Physical Activity Among Low Active Working Adults
Brief Title: A Video Chat Intervention for Enhancing Self-efficacy for Lifestyle Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Sean Mullen, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 19544
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Physical Activity; Self Efficacy; Working Adults
Keywords: leisure-time physical activity; adherence; working adults; motivation; social cognitive theory; telemedicine; teleconference; self-perceptions; self-confidence
MeSH Terms: conditions — Motor Activity | interventions — Work-Life Balance

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be blinded to the true purpose of the study. The investigators will be blinded to group assignment. The research assistants will be blinded to the true purpose of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efficacy for Lifestyle PA (Experimental): Three brief (10-minute) video chats during first three weeks of six weeks of lifestyle physical activity engagement providing information relative to outcome expectations (week 1), self-efficacy (week 2), and self-regulatory strategies (week 3) to enhance self-efficacy for lifestyle physical activity.
  Interventions: Behavioral: Efficacy for Lifestyle PA
- Efficacy for Work-life Balance (Active Comparator): Three brief (10-minute) video chats during first three weeks of six weeks of lifestyle physical activity engagement providing information relative to outcome expectations (week 1), self-efficacy (week 2), and self-regulatory strategies (week 3) to enhance self-efficacy for work-life balance.
  Interventions: Behavioral: Efficacy for Work-life Balance

INTERVENTIONS:
Behavioral: Efficacy for Lifestyle PA — The intervention group is asked to participate in three (10-minute) video chats during the first three weeks of six weeks of engaging in lifestyle physical activity. Participants in this group will receive information that addresses outcome expectations in week one (e.g. physical, social, and self-evaluative outcomes and intrinsic and extrinsic motives), self-efficacy in week two (e.g. the four efficacy sources: vicarious experiences, mastery experiences, social persuasion, and perceptions of physiological and affective responses to behavior), and self-regulatory strategies in week three (e.g. goal-setting, self-monitoring, and planning) for engaging in lifestyle physical activity.
  Other Names: intervention group
  Arms: Efficacy for Lifestyle PA
Behavioral: Efficacy for Work-life Balance — The time-matched control group is asked to participate in three (10-minute) video chats during the first three weeks of six weeks of engaging in lifestyle physical activity. Participants in this group will receive information that addresses outcome expectations in week one (e.g. physical, social, and self-evaluative outcomes and intrinsic and extrinsic motives), self-efficacy in week two (e.g. the four efficacy sources: vicarious experiences, mastery experiences, social persuasion, and perceptions of physiological and affective responses to behavior), and self-regulatory strategies in week three (e.g. goal-setting, self-monitoring, and planning) for work-life balance.
  Other Names: time-matched control group
  Arms: Efficacy for Work-life Balance

SUMMARY:
The purpose of this study is to evaluate the efficacy of three, brief (10-minute) theory-guided video chats for increasing self-efficacy for lifestyle physical activity versus a time-matched video chat comparison group designed to increase self-efficacy for work-life balance. Participants will include individuals who are low-active, full-time (>35 hours/week) working adults.

DETAILED DESCRIPTION:
Eligible participants will complete three brief (10-minute) video chats to promote self-efficacy during the first three weeks of engaging in lifestyle physical activity. Randomization will place participants into one of two groups: (1) Social Cognitive Theory-guided video chat or (2) time-matched video chat comparison group. Video chats will be delivered via the Google Duo smartphone app.

Baseline and follow-up assessments will consist of psycho-social questionnaires assessing constructs of the Social Cognitive Theory, affect, stress, and work-life balance. Physiological measures including heart rate will be assessed during a baseline treadmill assessment (to be completed in lab). All participants, regardless of group, will be asked to wear an activity tracker for the entirety of the study for assessing lifestyle physical activity. The comparison group will be asked to complete all baseline and follow-up assessments but will not receive information relative to lifestyle physical activity. The baseline assessments will take place with an academic research laboratory and weeks 2-7 will take place off outside of the lab.

ELIGIBILITY:
Inclusion Criteria:

* 25-64 years of age
* inactive (defined as not participating in exercise for 2 or more days per week for >30 minutes over the past 3-months)
* willing to be randomized to any condition
* owns iOs or Android smartphone

Exclusion Criteria:

* unable to speak or read English
* having a cognitive impairment (assessed via modified Telephone Interview for Cognitive Status [TICS]; score less than 21 will result in study exclusion)
* unable to exercise at moderate intensity level without causing or exacerbating a pre-existing condition which prevents participation in an exercise program

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Change in Self-efficacy for Lifestyle Physical Activity (SELPA) | Assessed at baseline, at week 2, 3, and 4, as well as end of study (beginning of week 8)
  The SELPA is a 6-item questionnaire that assesses beliefs in one's ability to engage in physical activity of one's own choosing to meet the physical activity guidelines. The SELPA is a modified version of the Lifestyle Efficacy Scale (McAuley, Hall, Motl, Wojcicki, White, Hu, & Doerksen, 2009). In this study, participants are asked to assess their confidence in their ability to accumulate five or more times per week at a moderate intensity, for at least 30 minutes for six weeks. Each question is based on a confidence scale ranging from 0% (not confident at all) to 100% (highly confident). The SELPA composite score is calculated by summing and averaging the six items, with higher scores representing greater self-efficacy for lifestyle physical activity.

SECONDARY OUTCOMES:
Lifestyle Physical Activity (subjective) | Assessed at baseline and at 6-week follow-up
  Lifestyle physical activity will be assessed via the Godin Leisure-Time Exercise Questionnaire (GLTEQ; Godin & Shephard, 1985), a brief, 4-item measure of physical activity that asks individuals to assess their current frequencies of engaging in strenuous, moderate, and light activities for at least 15 minutes per session during a typical week.Total weekly leisure activity is calculated by the equation: (9*strenuous) + (5*moderate) + (3*light). The second question assesses the frequency of weekly leisure-time activities that are done long enough for the individual to "work up a sweat."
Lifestyle Physical Activity (objective) | Assessed for entirety of 7-week study
  Lifestyle physical activity will be objectively measured using the Fitbit Charge 3 activity and sleep tracker. The Fitbit Charge 3 is a small device that measures all-day activity, distance, floors climbed, and sleep. The participants will be asked to wear the device for seven consecutive days (24 hours/day) prior to the brief in-person assessment and upon completion of the in-person assessment, all participants will be asked to wear the device for the entirety of the six weeks of the study period. Lifestyle physical activity will be assessed through "active minutes," or time spent in moderate-intensity activity.
Positive and Negative Feeling States | Assessed at week 1 (pre/post-treadmill assessment)
  The Feeling Scale (FS; Hardy & Rejeski, 1989), consists of a single-item assessing feelings of pleasure-displeasure, ranging from -5 (very bad) to +5 (very good). Participants are asked how the exercise makes them feel. The FS is scored based upon the number provided by the participant, with a possible range of -5 to +5, with higher scores indicating greater feelings experienced.
Anticipated Negative Affect | Assessed at week 1 (pre/post-treadmill assessment)
  Anticipated negative emotions will be assessed via the Anticipated Negative Affect Questionnaire (ANAQ; Wang, 2011). The ANAQ asks participants to anticipate how they may feel not regularly participating in physical activity. The ANAQ consists of 5 bi-polar items: "relaxed/tense," "not guilty/guilty," "no regret/regret," "not angry/angry," and "displeased/pleased." The ANAQ scale ranges from 1 to 7. Anticipated negative affect is scored based upon the number provided for each individual question, with higher scores indicating more negative emotions.
Forecasted Pleasure | Assessed at week 1 (pre/post-treadmill assessment)
  Forecasted pleasure will be assessed via one question "If you repeated the exercise session again, how do you think it would make you feel?" (Zenko et al., 2016). Responses are recorded by selecting from 15 empirically spaced anchors, ranging from -100 (most unpleasant imaginable) to +100 (most pleasant imaginable). Forecasted pleasure is scored based upon the number provided by the participant, with a possible range of -100 to +100, with higher scores indicating more pleasant, imaginable feelings.
Sedentary Behavior | Assessed at baseline and at 6-week follow-up
  The Sedentary Behavior Questionnaire (SBQ; Rosenberg et al., 2010) will be used to assess individual's self-reported sedentary behavior. The SBQ assesses the amount of time spent doing nine sedentary behaviors (watching television, playing computer/video games, sitting while listening to music, sitting and talking on the phone, doing paperwork or office work, sitting and reading, playing a musical instrument, doing arts and crafts, sitting and driving/riding in a car, bus, or train). The SBQ assesses sedentary time on a typical weekday and weekend day. Total sedentary behavior is calculated by recoding time reported into hours, then summing the total hours for all nine measures, for the weekday and weekend day. Weekly estimates are calculated by multiplying the weekday hours by (5) and the weekend day hours by (2), and summing together for total sedentary hours per week.
General Stress | Assessed at baseline and at 6-week follow-up
  General stress will be assessed via the Perceived Stress Scale (PSS; Cohen, Kamarck, & Mermelstein, 1983). The PSS is a 10-item questionnaire and scores are obtained by reverse scoring on four positive items and then summing across all items. Each question is based on a 5-point Likert scale, ranging from 0 (never) to 4 (very often). Higher scores indicates higher levels of general stress.
Job-related Stress | Assessed at baseline and at 6-week follow-up
  Job stress will be assessed via the Brief Job Stress Questionnaire (BJSQ; Kawada & Otsuka, 2011). The BJSQ is a 15-item scale that has 4 subscales: evaluation of job demand, job control, support, and degree of job satisfaction. Each question is based on a 4-point Likert scale, ranging from 1 (disagree) to 4 (agree). Each subscale is scored by summing the total items (reverse scoring the job demand subscale), with higher scores being indicative of lower job stress.
Exercise Planning and Scheduling | Assessed at baseline and at 6-week follow-up
  The Exercise Planning and Schedule Scale (EPSS; Rovniak, Anderson, Winett, & Stephens, 2002) is a 10-item questionnaire that assesses exercise scheduling and planning. Each question is based on a 5-point Likert scale, ranging from 1 (does not describe me) to 5 (describes me completely). The EPSS composite score is calculated by reverse-scoring items 2, 3, and 7 then summing and averaging the 10-items to create a composite score. Higher scores indicate more scheduling and planning done for exercise.
Physical Activity Self-regulation | Assessed at baseline and at 6-week follow-up
  The Physical Activity Self-regulation Scale (PASR-12; Umstattd et al., 2009) assesses the degree to which self-regulation strategies are used to support physical activity behavior. The PASR-12 is a 12-item questionnaire and the composite score is calculated by summing the 12-items. There are six subscales within the PASR-12 (calculated by summing the designated items): self-monitoring, goal-setting, social support, reinforcement, time management, and relapse prevention. Higher scores indicate greater strategy-use (either by subscale or composite score of total strategies used).
Self-efficacy to Regulate Work and Life | Assessed at baseline, at week 2, 3, and 4, as well as end of study (beginning of week 8)
  The Self-efficacy to Regulate Work and Life Questionnaire is a 5-item questionnaire that assesses how confident individuals are in regulating their work and non-work domains (Chan et al., 2016).The five items include: 1) "How confident are you in changing your lifestyle to achieve a good work-life balance?," 2) "How confident are you in finding out how to balance work and life?," 3) "How confident are you in achieving your ideal work-life balance?," 4) "How confident are you in implementing strategies to achieve work-life balance?," and 5) "How confident are you in inventing ways to balance your work and life?." Responses to all items are based on a scale ranging from 0 (cannot do at all) to 100 (highly certain can do). The composite score is calculated by summing and averaging the five items, with higher scores indicating that individuals are more confident in their abilities to cope with work-life challenges.
Outcome Expectancies for Exercise | Assessed at baseline and at 6-week follow-up
  The Multidimensional Outcome Expectancies for Exercise Scale (MOEES; Wójcicki, White, & McAuley, 2009) is a 15-item questionnaire that has three subscales: physical outcome expectancies, social outcome expectancies, and self-evaluative outcome expectancies. The MOEES assesses an individual's beliefs or expectations about the benefits of regular exercise. Each question is based on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). Each subscale is scored by summing the total items, with higher scores being indicative of higher outcome expectations for exercise.
Work-life Balance | Assessed at baseline and at 6-week follow-up
  The work-life balance scale (WLB-6; Gröpel & Kuhl, 2009) is a 6-item questionnaire that measures perceived sufficiency of time available for work and social life. Each question is based on a 6-point Likert scale, ranging from 1 (completely disagree) to 6 (completely agree). The WLB-6 is scored by reverse coding select items and summing the total items, with higher scores being indicative of high work-life balance.
Exercise Self-Schema | Assessed at baseline and at 6-week follow-up
  The Exercise Self-Schema Questionnaire (ESSQ; Kendzierski, 1988) was originally a 9-item scale. We are using a modified version which includes an additional item reflecting self-certainty ratings for each self-description item, as well as an extra question reflecting self-description, -importance, and -certainty with regard to "I am someone who will always be an exerciser" (Mullen, 2011). This version is a 12-item questionnaire and each question is based on an 11-point Likert Scale, ranging from 1 (does not describe me) to 11 (describes me). The ESSQ will be scored by summing and averaging the subscales (self-description, importance, certainty), with higher scores indicating greater exercise schema. Schematics can also be determined by categorizing responses to self-description and importance items that fall within the 8 to 11 range. In this study, change in self-schema will be assessed via changes in mean levels of the continuous variables rather than the dichotomous categorization.
Self-efficacy for Physical Activity | Assessed at baseline and at 6-week follow-up
  The Sources of Self-efficacy for Physical Activity (Warner et al., 2014) is an 18-item questionnaire that measures mastery experience, self-persuasion, verbal persuasion, vicarious experience, negative affect, and positive affect relative to physical activity. Each question is based on a 4-point Likert Scale, ranging from 1 (strongly disagree) to 4 (strongly agree). The questionnaire is scored by summing and averaging the subscales, with higher scores indicating greater use of self-efficacy sources.

OTHER OUTCOMES:
Overall Enjoyment with Physical Activity | Assessed at 6-week follow-up
  The Physical Activity Enjoyment Scale (PACES; Kendzierski & DeCarlo, 1991) is an 18-item questionnaire and items are based on a 7-point Likert scale, ranging from 1 (e.g. it makes me depressed) to 7 (e.g. it makes me happy). The PACES is scored by reverse coding items 1, 4, 5, 7, 9, 10, 11, 13, 14, 16, and 17 and then summing all of the items, with scores ranging from 7 to 126. Higher scores indicate greater physical activity enjoyment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tiffany Bullard, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Although this is not an NIH-funded study, we will update these records within 1 year of data collection per NIH guidelines.
Access Criteria: Data will be accessible on an open site (e.g. Open Science Framework https://osf.io/) with a request to interested parties to engage with the investigative team about any publication of these data in an effort to avoid redundancy. Appropriate authorship crediting investigators involved in the parent study conceptualization, and any consultation regarding data interpretation should be sought by any researchers interested in publishing these data.

REFERENCES:
- See also: Exercise, Technology, and Cognition Laboratory — http://exercisetechlab.com